CLINICAL TRIAL: NCT04855071
Title: Effectiveness and Safety of Non-ablative Radiofrequency in the Treatment of Pelvic Organ Prolapse and Its Associated Symptoms
Brief Title: Radiofrequency and Pelvic Organ Prolapse
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundació d'investigació Sanitària de les Illes Balears (Other Government)
Collaborators: University of the Balearic Islands (Other)
Responsible Party: Principal Investigator, Juan Carlos Fernández Domínguez, PhD, Fundació d'investigació Sanitària de les Illes Balears
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IB4459/21PS
Record Dates: First submitted 2021-03-10; First posted 2021-04-22 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Pelvic Organ Prolapse
Keywords: Radiofrequency Therapy; Pelvic floor muscle training; Quality of Life; Low Back Pain; Women; Safety
MeSH Terms: conditions — Pelvic Organ Prolapse; Low Back Pain

STUDY DESIGN:
Intervention Model Description: IG receives the usual intervention, which consists of performing exercises to balance the pelvis and their muscles and activation of the transverse abdominis and pelvic floor muscles and life habit advices plus the application of RF sessions.
  CG receives only the usual intervention. Sham RF sessions will be applied, using the same protocol as for the IG.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The women will be assigned to each of the study groups in an individualized random way, based on the table of random numbers generated prior to the start of the study through the EPIDAT v.4 software (Galicia, Spain). The randomization sequence will be kept hidden, through the use of sealed and opaque envelopes previously prepared by the main investigator of the project (JCFD) and which will be placed in a box available to the physiotherapists who perform each of the interventions.
  The allocation of women to the treatment groups will be blinded and also the blinding will be maintained in the analysis (evaluation of results), in such a way that in the data analysis only the groups will be identified.
  It is not possible to blind the physiotherapist professionals who perform the intervention (neither in the IG nor in the CG).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Active Comparator): The intervention will consist of supervised individualized sessions that will include application of exercises to balance the pelvis and their muscles, treatment of trigger points, teaching activation of the transverse abdominis with ultrasound biofeedback and teaching reflex activation exercises of the transverse abdominis and pelvic floor muscles in different body positions. In addition, standards of water, urination, food, defecation, postural hygiene and physical activity will be provided. It is also recommended different life habit advices related to tobacco use, constipation, etc.
  Furthemore, active RF will be applied intracavitary, in monopolar application, reaching a temperature between 42-45ºC in the tissues (according to the patient's tolerance), and with a power of 50% until the desired temperature is reached. It will be applied with a dose of approximately between 3-4 KJ depending on the application time (20 minutes / session).
  Interventions: Device: Non-ablative radiofrequency application; Other: Usual intervention
- Comparator group (Sham Comparator): The intervention will be the same that in IG (exercises to balance the pelvis and their muscles, etc) an also standards of water, urination, food, defecation, postural hygiene and physical activity for their generalization at home and life habit advices. The application of RF in the control group will follow the same application procedure as in the intervention group with the only difference that no parameter is applied to the RF device (in terms of temperature, power, frequency and dose); that is, it remains off for the entire duration of the session.
  Interventions: Other: Usual intervention

INTERVENTIONS:
Device: Non-ablative radiofrequency application — Non-ablative radiofrequency application will be applied with MJS intracavitary probe, in monopolar application, reaching a temperature between 42-45ºC in the tissues (according to the patient's tolerance), and with a power of 50% until the desired temperature is reached. It will be applied with a frequency that will be individualized according to the maximum level of energy absorption by the patient's tissues (between 0.8-1.2MHz) and with a dose of approximately between 3-4 KJ depending on the application time (20 minutes / session). In addition, they will be applied 1 session per week. The treatment will last 8 weeks.
  Other Names: Usual intervention
  Arms: Interventional group
Other: Usual intervention — The usual intervention will consist of supervised individualized sessions that will include application of exercises to balance the pelvis and their muscles, treatment of trigger points, teaching activation of the transverse abdominis with ultrasound biofeedback and teaching reflex activation exercises of the transverse abdominis and pelvic floor muscles in different body positions. In addition, standards of water, urination, food, defecation, postural hygiene and physical activity will be provided. It is also recommended different life habit advices related to tobacco use, constipation, etc.

SUMMARY:
Aim To compare the effectiveness of the application of non-ablative radiofrequency (RF) applied in combination with the usual treatment for the treatment of pelvic organ prolapse (POP) versus the usual treatment in lowering its severity.

The secondary objective is to compare the effectiveness of both interventions in the symptoms most commonly associated with POP (pelvic heaviness, bulging, and prolapse-related lumbar pain).

Design Randomized, double-blind clinical trial. Women between 18 and 75 years old with symptoms of vaginal prolapse, defined as "sensation of mass or lump" and / or "sensation of dragging in the vagina", and who also have the presence of POP diagnosed under clinical criteria and quantified using simplified POP-Q assessment.

All women with asymptomatic vaginal prolapse grade IV or less than GI of the cervix or less than or equal to GI of the anterior and / or posterior vaginal Wall (asymptomatic); presence of more than one vaginal prolapse, and also those women with chronic connective tissue diseases or who present some type of contraindication to the application of RF therapy, will be excluded from the study Methods The study will include 20 women in the intervention group and 20 women in the control group.

The women will be recruited from the patients who attend the Ketty Ruiz Pelviperineal Physiotherapy Clinic, which it´s specialized in treating pelvic floor dysfunctions.

Interventions The usual intervention will be applied to both groups of the study. It will consist of supervised individualized sessions (up to a maximum of 8 sessions) by physiotherapists who are part of the research team. They will include the application of exercises to balance the pelvis and the muscles related to it, treatment of the trigger points detected through the application of manual and / or instrumental techniques, teaching of the activation of the transverse abdominis with ultrasound biofeedback and teaching of reflex activation exercises of the transverse abdominis and pelvic floor muscles in different body positions.

The RF will be administered during the exercises of reflex activation of transversus abdominis and pelvic floor muscles on a stretcher (supine position). It will be applied intracavitary, in monopolar application, reaching a temperature between 42-45ºC in the tissues (according to the patient's tolerance), and with a power of 50% until the desired temperature is reached. It will be applied with a frequency that will be individualized according to the maximum level of energy absorption by the patient's tissues (between 0.8-1.2MHz) and with a dose of approximately between 3-4 KJ depending on the application time (20 minutes / session). In addition, they will be applied 1 session per week. The treatment will last 8 weeks.

The application of RF in the control group will follow the same application procedure as in the intervention group, but in this case, no type of parameter is applied to the RF device, ie, the device remains off for the entire duration of the session.

Variables:

For the measurement of the main variable of the study, the simplified POP-Q will be used, considered the "gold standard" for the classification of POP. To measure the secondary variables of the study, the Pelvic Organ Prolapse Symptom Score (POP-SS) questionnaire will be used to assess the symptoms of pelvic bulging and / or heaviness; a visual analog scale (VAS) for the intensity of lumbar pain related to prolapse, the Prolapse Quality of Life (P-QOL) questionnaire for measuring the quality of life related to vaginal prolapse and finally structured interviews will be conducted with all study subjects throughout the duration of the study to assess the safety of the intervention The immediate effect (ie, at the end of the 1st treatment session) in the quantitative assessment of prolapse and the short-term effects (i.e. 1 week after the last face-to-face treatment session) and medium (at 3 and 6 months after end of treatment) and long-term effects (at 12 months after finishing treatment) in all study variables will be evaluated.

Statistical analysis and ethical aspects It will be carried out using the SPSS 25.0 statistical package. This project is in process of being approved by the Research Ethics Committee (CEI) of the Balearic Islands (IB 4459/21 PS).

DETAILED DESCRIPTION:
Effectiveness and safety of non-ablative radiofrequency in the treatment of pelvic organ prolapse and its associated symptoms OBJECTIVES Primary To compare the effectiveness of application of non-ablative radiofrequency applied in combination with the usual treatment versus usual treatment for the treatment of pelvic organ prolapse (POP) - specifically in the reduction of vaginal prolapses.

Secondary To compare the effectiveness of both interventions in the symptoms most commonly associated with vaginal prolapse (pelvic heaviness, bulging, and POP-related low back pain).

Specific

* To analyze the prevalence of symptoms associated with vaginal prolapse depending on the stage of POP.
* Compare the effectiveness depending on the location of prolapse: anterior vaginal wall, posterior vaginal wall or vaginal vault.
* Compare the effectiveness according to the degree of prolapse (stages extracted from the simplified POP-Q: I, IIA, IIB and III).
* Compare the effectiveness based on age.
* Evaluate the relationship of vaginal prolapse symptoms with the location and severity of vaginal prolapse, respectively in the anterior, posterior and apex wall (Ba, Bp and C).
* Evaluate the immediate effect of RF application on the stage of prolapse.
* Estimate the effect of both interventions (usual treatment vs usual treatment with active RF), at the end of the 1st treatment session and after finishing the treatment: short (1 week after the last session), medium (at 3 and 6 months post-intervention) and long-term (at 12 months post-intervention) on the quantitative assessment of POP and the most commonly associated symptoms.
* Evaluate the safety of the RF technique (presence of adverse events)

METHODOLOGY DESIGN Double-blind clinical trial with two interventions: usual treatment for POP versus the usual treatment including application of RF. These interventions are randomly assigned. The full follow-up period is 12 months. The study design conforms to the recommendations of the Consolidated Standards of Reporting Trials (CONSORT) for Statement to Randomized Trials of Nonpharmacological Treatment.

SAMPLE SELECTION CRITERIA

1. Subject inclusion criteria

   * Women between 18 and 75 years old.
   * Women who state symptoms of vaginal prolapse, defined as "sensation of mass or lump" and / or "sensation of dragging in the vagina" and who also have the presence of POP; i.e. descent of one of the anterior, posterior or uterus vaginal walls (cervix) diagnosed under clinical criteria and quantified using the simplified POP-Q assessment system.
2. Criteria for exclusion of subjects

   * Prolapse vaginal GIV (according to clinical stage evaluated by POP-Q -Pelvic Organ Prolapse Quantification-).
   * Presence of more than one POP
   * Asymptomatic vaginal prolapse grade IV or less than GI of the cervix or less than or equal to GI of the anterior and / or posterior vaginal Wall
   * Women with chronic connective tissue diseases
   * Women who present contraindication to the application of RF therapy such as: pregnancy, metallic prostheses within the electric field, decompensated arteriopathies, malignant neoplasms, active infectious processes, pacemakers, loss of thermal sensitivity,….
3. Study withdrawal criteria

   * Revocation of informed consent
   * Presence of severe adverse effects derived from RF treatment

   RECRUITMENT The study will be carried out by the University of the Balearic Islands. The women will be recruited from the patients who attend the Ketty Ruiz Pelviperineal Physiotherapy Clinic, which it´s specialized in treating pelvic floor dysfunction.

   The control group (CG) will receive the usual intervention (described later) plus the "sham RF" application, that is, not active; while the intervention group (IG) will receive the same usual intervention that is provided to the CG subjects plus the application of active RF in the parameters that are considered most appropriate for the approach of this kind of dysfunction (described later) The application of sham-RF will allow, on the one hand, to blind women who have never received RF treatment and will also allow the assessment of placebo effect of the RF application itself.

   The interventions will be carried out by members of the work team, made up of 3 physiotherapists specialized in pelvic floor physiotherapy (KRL, ELlF, MAQ). The homogeneity of the so-called "usual intervention" will be ensured because all the physiotherapists who work in the clinic where the intervention is carried out (KRL, ELlF, MAQ) use the same work protocol for the treatment of POPs. In addition, for the application of RF (sham or active) a standardized protocol will be followed, to remove differences in RF application that may influence the results obtained.

   INTERVENTIONS USUAL INTERVENTION The usual intervention begins with a physical examination that includes the assessment of the strength of pelvic floor muscles (PFM) using the PERFECT method, assessment of tone of PFM to rule out hypertonia, ultrasound evaluation of the abdominal-perineal synergies and electromyographic assessment (by surface EMG) of pelvic floor and internal oblique muscles.

   The intervention will consist of supervised individualized sessions (up to a maximum of 8 sessions) by physiotherapists who are part of the research team. They will include the application of exercises to balance the pelvis and the muscles related to it, treatment of the trigger points detected through the application of manual and / or instrumental techniques, teaching of the activation of the transverse abdominis with ultrasound biofeedback and teaching of reflex activation exercises of the transverse abdominis and pelvic floor muscles in different body positions. If PFM strength is less than 3 on modified Oxford scale, intravaginal electrotherapy (muscle electrostimulation) will be applied. All treatment techniques will be adapted individually based on the results obtained in the previous physical examination process.

   In addition to the supervised sessions, the patient is given an exercise sheet that includes reflex postural activation of transversus abdominis muscle and PFM by means of slowed exhalation to be carried out daily (even after the supervised treatment sessions have ended).

   In addition, within the "usual intervention", standards of water, urination, food, defecation, postural hygiene and physical activity for their generalization at home are given to all women. They are provided with information on voiding and defecation physiology and the importance of maintainance proper habits in each of these fields.

   It is recommended the reduction or even avoidance of tobacco consumption, limit caffeine intake, eat a balanced diet according to the Harvard dish to avoid constipation, avoid weight gain or recommend to lose weight in case of overweight and avoid lifting weight, as well as playing high-impact sports.

   Patients who also present constipation (according to Rome IV criteria) are instructed in proper habits to go to the bathroom, avoiding the push / tension of the pelvic floor. Finally, patients with loss of abdominoperineal anticipation synergies (through ultrasound evaluation) are taught the knack maneuver before and during any task that involves an increase in intra-abdominal pressure.

   RADIO FREQUENCY IG: active RF The active RF will be administered during the exercises of reflex activation of transversus abdominis and pelvic floor muscles on a stretcher (supine position).

   It will be applied intracavitary, in monopolar application, reaching a temperature between 42-45ºC in the tissues (according to the patient's tolerance), and with a power of 50% until the desired temperature is reached. It will be applied with a frequency that will be individualized according to the maximum level of energy absorption by the patient's tissues (between 0.8-1.2MHz) and with a dose of approximately between 3-4 KJ depending on the application time (20 minutes / session). In addition, they will be applied 1 session per week. The treatment will last 8 weeks.

   CG: sham RF The application of RF in the control group will follow the same application procedure as in the intervention group i. e. it will be applied during the exercises of reflex activation of transversus abdominis and pelvic floor muscles on a stretcher (supine position) and with the same technical execution (including technical application and duration of session, weekly frequency and total number of sessions). The only difference will be that in the CG subjects, no parameter is applied to the RF device (in terms of temperature, power, frequency and dose); that is, it remains off for the entire duration of the session.

   FOLLOW-UP The immediate and the short, medium and long term effects will be assessed
   * Inmediate effect: the immediate effect of both treatments will be compared ("usual intervention" plus " sham RF " vs "usual intervention" plus "active RF") in the quantitative assessment of prolapse (through simplified POP-Q).
   * Short term: the effect of both treatments at the end of the RF sessions (1 week after the last session) will be compared both in the quantitative assessment of prolapse (through simplified POP-Q) and in the symptoms most commonly associated with vaginal prolapses: pelvic heaviness, bulging and low pelvic-lumbar pain related to POP (through the measurement instruments described in the section "Outcomes and measurement instruments"). The potential adverse events of RF in both groups (CG and IG) will also be assessed.
   * Medium term: three and six months after the end of the treatment, the effect of both treatments will be compared on the previously mentioned variables.
   * Long-term: twelve months after the end of the treatment, the effect of both treatments will be compared on the variables mentioned above.

   OUTCOMES AND MEASUREMENT INSTRUMENTS Main variable Degree of prolapse through the simplified POP-Q (Parekh et al. 2011; Swift et al. 2006). This standardized prolapse assessment method has excellent inter and intra observer reliability, as well as a significant association between assessments using the POP-Q and the simplified POP-Q itself (Manonai et al., 2011). This instrument is internationally recognized, being considered the "gold standard" for prolapse classification (Hall et al., 1996).

   For this, measurements that allow the quantitative description of the position of the pelvic organs (i.e. the numerical values in cm of the various vaginal segments) will be used (Bump 2014; Bump et al, 1996), specifically:
   * Anterior vaginal segment: called point Ba (estimated around 3 cm proximal to the hymenal caruncles)
   * Posterior vaginal segment: called point Bp (estimated around 3 cm proximal to the hymenal caruncles)
   * Cervix: called point C
   * Posterior apex / fornix: called point D

   To measure these points, the subject is placed in a standardized dorsal lithotomy position (90º hip and knee flexion and with leg support on the gynecological stretcher), From there, the subject is asked to push hard, performing a standardized maximum Valsalva maneuver with a minimum of 5 s in duration (Orejuela et al., 2012), closing the mouth while pressing out as if the individual is straining to defecate (in order to demonstrate the maximum descent of the pelvic organs). A mirror is used to confirm the correlation of physical findings with the study participant's medical history (Manonai et al. 2016).

   Measurements will be made using a calliper, an hysterometer and a half leaflet of a Collin-type speculum following the procedure described by Busquets et al. (Busquets et al., 2009).

   In addition, it will also be included the measurement of:
   * Degree of prolapse (according to the simplified POP-Q classification): I, IIa, IIb, III and IV.
   * Prolapse location: anterior wall, posterior wall, cervix ("diagnosed" by ultrasound and physical examination) (Dietz & Mann, 2014; Dietz, 2019).

   Measurement standardization procedure To ensure that all measurements are carried out equally by the members of the work team, made up of 3 physiotherapists specialized in pelvic floor physiotherapy (KRL, ELlF, MAQ), a training activity will be carried out by the principal investigator. Furthermore, a pilot test to verify the intra- and inter-examiner reliability of the measurements with the POP-Q will be carried out.

   Secondary variables A. Related to the effectiveness of the intervention Symptoms of POP (vaginal prolapse)

   Measurement of the most frequent symptoms derived from vaginal prolapse:

   -Bulging It is defined as the sensation of bulging or that something is descending through the vaginal introitus. The woman claims that she notices a lump by direct palpation or that she sees it with the help of a mirror (Haylen et al., 2016).

   This symptom is considered prolapse-specific and correlates with the severity of the prolapse (Jelovsek et al., 2007, Ghetti et al., 2005).

   -Pelvic heaviness It is defined as the feeling of heaviness, pressure or a dragging sensation (pain or discomfort) in the suprapubic or pelvic area (Haylen et al., 2016).

   To measure prolapse symptoms, the Pelvic Organ Prolapse Symptom Score (POP-SS) questionnaire will be used in its Spanish version. It presents an adequate internal consistency with a Cronbach's alpha coefficient> 0.7. It has adequate validity to measure the symptoms of prolapse and correct sensitivity to change. It is especially important in scales that measure the effectiveness of interventions for the treatment of prolapse (Hagen et al., 2009).

   -Low back pain - related to POP- It is defined as a complaint of low back or sacrum pain (or quite similar to menstruation pain) temporarily associated with vaginal prolapse and that is relieved when the prolapse is reduced.

   It will be assessed using a visual analog scale (VAS). This scale allows one-dimensional assessment of pain intensity to be measured in a horizontal line of 100 mm, in which participants are asked to indicate the mean intensity of pain they feel, ranging from 0 mm (no pain) to 100 mm (the greatest pain imaginable). It is a simple, valid, reliable and reproducible method (Thong et al., 2018; Eizaga & García, 2015).

   Quality of life To measure quality of life related to prolapse symptoms, the Spanish validated version (Flores-Espinoza et al., 2015) of the Prolapse Quality of Life (P-QOL) questionnaire (Digesu et al., 2005) will be used. It shows an excellent content validity (CVI = 0.9), adequate construct validity concerned to its association with the severity of urogenital and intestinal symptoms (discriminative validity), and with respect to its correlation with the POP stages assessed by the POP- Q in the domains of "impact of prolapse", "personal relationships", "emotions" and "measures of severity". It also presents adequate internal consistency, with Cronbach's alpha values higher than 0.70 in all dimensions except for "severity measures".

   Satisfaction with treatment (Sodré et al. 2019) For the subjective evaluation of satisfaction with the treatment technique used, a 5-point Likert scale will be used: 1- very dissatisfactory, 2- dissatisfactory, 3- neutral, 4- satisfied, 5-very satisfied

   B. Basal
   * Age
   * Weight
   * Height
   * Waist circumference
   * Menopause (yes / no / presence of perimenopausal symptoms)
   * Use of hormone replacement therapy (in menopausal women)
   * Hysterectomy: total or subtotal
   * Women who have had previous surgeries for POP: type of intervention
   * Women who have had previous surgeries for incontinence: type of intervention
   * Consumption of hormonal contraceptive drugs (oral, contraceptive adhesive, vaginal ring, injectable contraceptive, contraceptive implant, other: to be specified)

   Obstetric history
   * Date of last delivery
   * Number of deliveries
   * Type of delivery (of each delivery): vaginal, instrumental, caesarean section
   * Episiotomy

   If the woman is in immediate postpartum (<6 months):
   * Current breastfeeding (yes / no / mixed)
   * Presence of POP diagnosed prior to the current pregnancy (yes / no)

   C. Related to the safety of the intervention Information about the safety of the intervention will be collected through interviews with the study subjects.

   All adverse events (AE) that occur from the beginning of the treatment procedure until the end of the study will be recorded by each of the intervening physiotherapists.

   For each AE, the description, start date, severity, duration and relationship with the treatment will be recorded. All AEs will be followed until they decline or, in the case of permanent damage, until the AEs stabilize and the overall clinical outcome is determined.

   It is also collected if the subjects had to discontinue the treatment, if they had to discontinue any session or if they had to stop the application of RF at some point during the course of treatment and their reason / s (Sodré et al. 2019).

   The relationship of the EA with the treatment will be determined by the IP of the project (JCFD) using the following classifications: related, possibly related, unknown and unrelated.

   Tamaño muestral:

   Sample size:

   The sample size for independent means with respect to both the CG and IG measurements has been obtained. Considering a bilateral contrast accepting an alpha risk of 0.05 and a beta risk of 0.20 and assuming a change in the main variable of the study, i.e. in the position of the pelvic organs of at least 15 mm, regardless of the vaginal segment (point Ba, Bp, C or D), a minimum total of 20 subjects in each group will be required for a total of 40 subjects, estimating a loss to follow-up rate of 20%.

   Randomization:

   The women will be assigned to each of the study groups in an individualized random way, based on the table of random numbers generated prior to the start of the study through the EPIDAT v.4 software (Galicia, Spain). The randomization sequence will be kept hidden, through the use of sealed and opaque envelopes previously prepared by the main investigator of the project (JCFD) and which will be placed in a box available to the physiotherapists who perform each of the interventions.

   Blinding It is not possible to blind the physiotherapist professionals who perform the intervention (neither in the IG nor in the CG).

   However, the allocation of women to the treatment groups will be blinded and also the blinding will be maintained in the analysis (evaluation of results), in such a way that in the data analysis only the groups will be identified.

   Statistical analysis A descriptive analysis of all variables, both categorical and quantitative, will be carried out, with frequency and percentage for categorial, and Exploratory Data Analysis (AED) for the latter; as well as the Shapiro-Wilk normality tests to establish compliance or not with the statistical assumptions of the parametric analysis. Shapiro-Wilk normality tests will be performed to establish compliance with the statistical assumptions for the parametric analysis.

   The differences in the baseline values between both study groups will be performed using parametric (Student's t-test for independent samples) or non-parametric (U-Mann Whitney) tests depending on the results of the goodness-of-fit tests. In case of statistically significant differences between the groups in the baseline measurements, the pre-intervention values will be included as a potential covariate (analysis of covariance) to adjust the effect.

   For the comparison between the pre and post intervention phases (at the end of the intervention, 3 months, 6 months and 12 months) in each study group with respect to the main and secondary variables related to both the effectiveness of the intervention and the quality of life, Student's t test for independent samples or the U-Mann Whitney test will be used. The effect size will be estimated using Cohen's d and the 95% confidence interval of the difference of the pre-post means in the study variables mentioned above.

   An analysis of the variance of repeated measures of two factors will be carried out using time (pre and post-1 - at the end of the intervention and post 2- at 3 months, post 3- at 6 months and post 4 - at 12 months) and the treatment group (control group vs. intervention).

   To check the immediate effect (after the 1st session) of the application of RF in the IG, an analysis for within-subject measurements using the Student's t test for paired means or the Wilcoxon test was performed. The effect size will also be estimated using Cohen's d and the 95% confidence interval to check the magnitude of the differences, if required.

   Data will be analyzed and processed using the SPSS v.25 statistical package. Ethical aspects The study will have the approval of the Committee of Ethics and Clinical Research (CEI) of the Balearic Islands (in process).

   All subjects in the study must be informed, and if they agree to participate, sign the informed consent.

   In the event that as a result of the treatment in the IG, significant results are obtained in relation to the variables studied, the research team undertakes to offer the same treatment and under the same conditions to the subjects randomly assigned to the GC, once the study period is over.

   Boutron I., Moher D., Altman DG., Schulz KF., Ravaud P.,& CONSORT Group. Extending the CONSORT statement to randomized trials of nonpharmacologic treatment: explanation and elaboration. Ann Intern Med. 2008;148(4):295-309. doi: 10.7326/0003-4819-148-4-200802190-00008.

   Bump RC. The POP-Q system: two decades of progress and debate. Int Urogynecol J. 2014;25(4):441-3. doi: 10.1007/s00192-013-2262-0 Bump RC, Mattiasson A, Bø K, Brubaker LP, DeLancey JO, Klarskov P, et al. The standardization of terminology of female pelvic organ prolapse and pelvic floor dysfunction. Am J Obstet Gynecol. 1996;175(1):10-7. doi: 10.1016/s0002-9378(96)70243-0.

   Busquets M., Castillo F., Bravo S., & Contreras D. Uso del sistema POPQ para la clasificación de los prolapsos: hospital parroquial de San Bernardo. Rev. Chil. Obstet. Ginecol. 2009;74(1):4-10. doi: 10.4067/S0717-75262009000100002 Dietz HP. Ultrasound in the assessment of pelvic organ prolapse. Best Pract Res Clin Obstet Gynaecol. 2019 Jan;54:12-30. doi: 10.1016/j.bpobgyn.2018.06.006. Epub 2018 Jun 28.

   Dietz HP., & Mann KP. What is clinically relevant prolapse? An attempt at defining cutoffs for the clinical assessment of pelvic organ descent. Int Urogynecol J. 2014;25:451-455. doi:10.1007/s00192-013-2307-4 Dietz HP., & Mann KP. What is clinically relevant prolapse? An attempt at defining cutoffs for the clinical assessment of pelvic organ descent. Int Urogynecol J. 2014;25:451-455. doi:10.1007/s00192-013-2307-4 Digesu GA., Khullar V., Cardozo L., Robinson D., & Salvatore S. P-QOL: a validated questionnaire to assess the symptoms and quality of life of women with urogenital prolapse. Int Urogynecol J Pelvic Floor Dysfunct. 2005;16(3):176-81; discussion 181. doi: 10.1007/s00192-004-1225-x.

   Eizaga R., & García M. Escalas de Valoración de Dolor. 2015. Available from: https://www.researchgate.net/publication/321462394_Escalas_de_Valoracion_de_Dolor Flores-Espinoza C., Araya AX., Pizarro-Berdichevsky J., Santos V., Ferrer M., Garin O., et al. Validation of the Spanish-language version of the Prolapse Quality of Life questionnaire in Chilean women. Int Urogynecol J. 2015;26(1):123-30. doi: 10.1007/s00192-014-2484-9 Ghetti C., Gregory WT., Edwards SR., Otto LN., & Clark AL. Pelvic organ descent and symptoms of pelvic floor disorders. Am J Obstet Gynecol. 2005;193(1):53-7. doi:10.1016/j.ajog.2004.12.004 Hagen S., Glazener C., Sinclair L., Stark D., & Bugge C. (2009). Psychometric properties of the pelvic organ prolapse symptom score. BJOG. 2009;116(1):25-31. doi:10.1111/j.1471-0528.2008.01903.x Haylen BT, Maher CF, Barber MD, Camargo S, Dandolu V, Digesu A, et al. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic organ prolapse (POP). Int Urogynecol J. 2016;27(4):655-84. doi: 10.1007/s00192-016-3003-y Hall AF., Theofrastous JP., Cundiff GW., Harris RL., Hamilton LF., Swift SE, et al.. (1996). Interobserver and intraobserver reliability of the proposed International Continence Society, Society of Gynecologic Surgeons, and American Urogynecologic Society pelvic organ prolapse classification system. Am J Obstet Gynecol. 1996;175(6): 1467-70; discussion 1470-1. doi:10.1016/s0002-9378(96)70091-1 Jelovsek JE., Maher C., & Barber M. D. Pelvic organ prolapse. Lancet 2007;369(9566): 1027-38. doi: 10.1016/S0140-6736(07)60462-0 Manonai J., Wattanayingcharoenchai R. Relationship between pelvic floor symptoms and POP-Q measurements. Neurourol Urodyn. 2016 Aug;35(6):724-7. doi: 10.1002/nau.22786. Epub 2015 Apr 28.

   Manonai J., Mouritsen L., Palma P., Contreras-Ortiz O., Korte JE., & Swift S. The inter-system association between the simplified pelvic organ prolapse quantification system (S-POP) and the standard pelvic organ prolapse quantification system (POPQ) in describing pelvic organ prolapse. Int Urogynecol J. 2011;22(3):347-52. doi: 10.1007/s00192-010-1286-y. Epub 2010 Oct 9.

   Orejuela FJ., Shek KL., Dietz HP. The time factor in the assessment of prolapse and levator ballooning. Int Urogynecol J. 2012 Feb;23(2):175-8. doi: 10.1007/s00192-011-1533-x.

   Parekh M., Swift S., Lemos N., Iskander M., Freeman B., Arunkalaivanan AS., et al. Multicenter inter-examiner agreement trial for the validation of simplified POPQ system. Int Urogynecol J. 2011;22(6):645-50. doi: 10.1007/s00192-011-1395-2.

   Sodré DSM., Sodré PRS., Brasil C., Teles A., Dória M., Café LE., et al. New concept for treating urinary incontinence after radical prostatectomy with radiofrequency: phase 1 clinical trial. Lasers Med Sci. 2019;34(9):1865-71. doi: 10.1007/s10103-019-02784-7 Swift S, Morris S, McKinnie V, Freeman R, Petri E, Scotti RJ, et al. Validation of a simplified technique for using the POPQ pelvic organ prolapse classification system. Int Urogynecol J Pelvic Floor Dysfunct. 2006;17(6):615-20. doi: 10.1007/s00192-006-0076-z.

   Thong ISK., Jensen MP., Miró J., & Tan G. The validity of pain intensity measures: What do the NRS, VAS, VRS, and FPS-R measure? Scand J Pain. 2018;18(1):99-107. doi: 10.1515/sjpain-2018-0012 Toozs-Hobson P., Swift S. POP-Q stage I prolapse: is it time to alter our terminology? Int Urogynecol J. 2014;25(4):445-6. doi: 10.1007/s00192-013-2260-2

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 75 years old.
* Women who state symptoms of vaginal prolapse, defined as "sensation of mass or lump" and / or "sensation of dragging in the vagina" and who also have the presence of POP; i.e. descent of one of the anterior, posterior or uterus vaginal walls (cervix) diagnosed under clinical criteria and quantified using the simplified POP-Q assessment system.

Exclusion Criteria:

* Prolapse vaginal GIV (according to clinical stage evaluated by POP-Q -Pelvic Organ Prolapse Quantification-).
* Presence of more than one POP
* Asymptomatic vaginal prolapse grade IV or less than GI of the cervix or less than or equal to GI of the anterior and / or posterior vaginal Wall
* Women with chronic connective tissue diseases
* Women who present contraindication to the application of RF therapy such as: pregnancy, metallic prostheses within the electric field, decompensated arteriopathies, malignant neoplasms, active infectious processes, pacemakers, loss of thermal sensitivity,….
* Revocation of informed consent

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-04-23 (Estimated); Primary Completion 2022-10-23 (Estimated); Study Completion 2022-10-23 (Estimated)

PRIMARY OUTCOMES:
Change in degree of prolapse | Change from baseline degree of prolapse at the end of the first treatment session, at 9th week and at 3rd, 6th and 12th months, post treatment
  Quantitative description of the position of the pelvic organs through simplified POP-Q

SECONDARY OUTCOMES:
Changes in prolapse symptoms: bulging, pelvic heaviness and low back pain - related to POP- | Change from baseline in prolapse symptoms at 9 weeks and 3, 6 and 12 months post treatment
  Bulging: sensation of bulging or that something is descending through the vaginal introitus evaluated through Pelvic heaviness: feeling of heaviness, pressure or a dragging sensation (pain or discomfort) in the suprapubic or pelvic area evaluated.
  Both symptoms will be evaluated through the Pelvic Organ Prolapse Symptom Score (POP-SS) questionnaire in its Spanish versión.
  Low back pain - related to POP- : complaint of low back or sacrum pain (or quite similar to menstruation pain) temporarily associated with vaginal prolapse and that is relieved when the prolapse is reduced evaluated through a visual analog scale (VAS).
Changes in quality of life | Change from baseline in prolapse symptoms at 9 weeks and 3, 6 and 12 months post treatment
  To measure quality of life related to prolapse symptoms through the Spanish validated version of the Prolapse Quality of Life (P-QOL) questionnaire
Satisfaction with treatment | 12 months post treatment
  Subjective evaluation of satisfaction with the treatment technique used thrneutral, 4- satisfied, 5-very satisfied.

OTHER OUTCOMES:
Safety of RF intervention | Throughout the whole intervention
  Information about the safety of the intervention will be collected through interviews with the study subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Ketty K Ruiz-López, BSc, Study Director — Centro de fisioterapia pelviperineal Ketty Ruiz

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Boutron I., Moher D., Altman DG., Schulz KF., Ravaud P.,& CONSORT Group. Extending the CONSORT statement to randomized trials of nonpharmacologic treatment: explanation and elaboration. Ann Intern Med. 2008;148(4):295-309. — https://pubmed.ncbi.nlm.nih.gov/18283207/
- See also: Bump RC. The POP-Q system: two decades of progress and debate. Int Urogynecol J. 2014;25(4):441-3. — https://pubmed.ncbi.nlm.nih.gov/24504065/
- See also: Bump RC, Mattiasson A, Bø K, Brubaker LP, DeLancey JO, Klarskov P, et al. The standardization of terminology of female pelvic organ prolapse and pelvic floor dysfunction. Am J Obstet Gynecol. 1996;175(1):10-7. — https://pubmed.ncbi.nlm.nih.gov/8694033/
- See also: Busquets M., Castillo F., Bravo S., & Contreras D. Uso del sistema POPQ para la clasificación de los prolapsos: hospital parroquial de San Bernardo. Rev. Chil. Obstet. Ginecol. 2009;74(1):4-10. — https://scielo.conicyt.cl/scielo.php?script=sci_abstract&pid=S0717-75262009000100002&lng=pt&nrm=iso
- See also: Dietz HP. Ultrasound in the assessment of pelvic organ prolapse. Best Pract Res Clin Obstet Gynaecol. 2019 Jan;54:12-30. — https://pubmed.ncbi.nlm.nih.gov/30082146/
- See also: Dietz HP., & Mann KP. What is clinically relevant prolapse? An attempt at defining cutoffs for the clinical assessment of pelvic organ descent. Int Urogynecol J. 2014;25:451-455. doi:10.1007/s00192-013-2307-4 — https://pubmed.ncbi.nlm.nih.gov/24504066/
- See also: Digesu GA., Khullar V., Cardozo L., Robinson D., & Salvatore S. P-QOL: a validated questionnaire to assess the symptoms and quality of life of women with urogenital prolapse. Int Urogynecol J Pelvic Floor Dysfunct. 2005;16(3):176-81; discussion 181. doi: — https://pubmed.ncbi.nlm.nih.gov/15875234/
- See also: Eizaga R., & García M. Escalas de Valoración de Dolor. 2015. — https://www.researchgate.net/publication/321462394_Escalas_de_Valoracion_de_Dolor
- See also: Flores-Espinoza C., Araya AX., Pizarro-Berdichevsky J., Santos V., Ferrer M., Garin O., et al. Validation of the Spanish-language version of the Prolapse Quality of Life questionnaire in Chilean women. — http://repositorio.uchile.cl/bitstream/handle/2250/133237/Validation-of-the-Spanish-language-version-of-the-Prolapse-Quality.pdf?sequence=1
- See also: Ghetti C., Gregory WT., Edwards SR., Otto LN., & Clark AL. Pelvic organ descent and symptoms of pelvic floor disorders. Am J Obstet Gynecol. 2005;193(1):53-7. doi:10.1016/j.ajog.2004.12.004 — https://pubmed.ncbi.nlm.nih.gov/16021058/
- See also: Hagen S., Glazener C., Sinclair L., Stark D., & Bugge C. (2009). Psychometric properties of the pelvic organ prolapse symptom score. BJOG. 2009;116(1):25-31. doi:10.1111/j.1471-0528.2008.01903.x — https://pubmed.ncbi.nlm.nih.gov/18947342/
- See also: Haylen BT, Maher CF, Barber MD, Camargo S, Dandolu V, Digesu A, et al. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic organ prolapse (POP). — https://pubmed.ncbi.nlm.nih.gov/26755051/
- See also: Interobserver and intraobserver reliability of the proposed International Continence Society, Society of Gynecologic Surgeons, and American Urogynecologic Society — https://pubmed.ncbi.nlm.nih.gov/8987926/
- See also: Jelovsek JE., Maher C., & Barber M. D. Pelvic organ prolapse. Lancet 2007;369(9566): 1027-38. — https://pubmed.ncbi.nlm.nih.gov/17382829/
- See also: Manonai J., Wattanayingcharoenchai R. Relationship between pelvic floor symptoms and POP-Q measurements. Neurourol Urodyn. 2016 Aug;35(6):724-7. doi: 10.1002/nau.22786. Epub 2015 Apr 28. — https://pubmed.ncbi.nlm.nih.gov/25919311/
- See also: The inter-system association between the simplified pelvic organ prolapse quantification system (S-POP) and the standard pelvic organ prolapse quantification system (POPQ) in describing pelvic organ prolapse — https://pubmed.ncbi.nlm.nih.gov/20936258/
- See also: Orejuela FJ., Shek KL., Dietz HP. The time factor in the assessment of prolapse and levator ballooning. Int Urogynecol J. 2012 Feb;23(2):175-8. — https://pubmed.ncbi.nlm.nih.gov/21887550/
- See also: Parekh M., Swift S., Lemos N., Iskander M., Freeman B., Arunkalaivanan AS., et al. Multicenter inter-examiner agreement trial for the validation of simplified POPQ system. Int Urogynecol J. 2011;22(6):645-50. — https://www.researchgate.net/publication/50832721_Multicenter_inter-examiner_agreement_trial_for_the_validation_of_simplified_POPQ_system
- See also: Validation of a simplified technique for using the POPQ pelvic organ prolapse classification system. Int Urogynecol J Pelvic Floor Dysfunct. 2006;17(6):615-20. — https://pubmed.ncbi.nlm.nih.gov/16598414/
- See also: Thong ISK., Jensen MP., Miró J., & Tan G. The validity of pain intensity measures: What do the NRS, VAS, VRS, and FPS-R measure? Scand J Pain. 2018;18(1):99-107. doi: 10.1515/sjpain-2018-0012 — https://pubmed.ncbi.nlm.nih.gov/29794282/
- See also: Toozs-Hobson P., Swift S. POP-Q stage I prolapse: is it time to alter our terminology? Int Urogynecol J. 2014;25(4):445-6. doi: 10.1007/s00192-013-2260-2v — https://pubmed.ncbi.nlm.nih.gov/24504064/